CLINICAL TRIAL: NCT07340099
Title: Community-Based Participatory Research to Study Church Implementation of an Evidence-Based Social Support Intervention to Increase Physical Activity Among Older African American Adults
Brief Title: Church Implementation of a Social Support Intervention to Increase Physical Activity in Older African American Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sara Wilcox, Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00138947; U48DP006780 (NIH)
Record Dates: First submitted 2025-12-22; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants; Chronic Diseases in Older Adults; Chronic Disease Prevention
Keywords: physical activity; walking; health promotion; chronic disease prevention; older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Walk Your Heart to Health program
  Interventions: Behavioral: Walk Your Heart to Health

INTERVENTIONS:
Behavioral: Walk Your Heart to Health — 32-week walking intervention delivered by church committees

SUMMARY:
Many effective interventions or programs are never put into practice. This quasi-experimental study will partner with AME churches in two areas of South Carolina to study how an evidence-based program is put into place by the church. The program, Walk Your Heart to Health, will include training in how churches can modify their practices to support physical activity and healthy eating. Over the five-year study, the investgiators will examine factors that predict the success of putting the program into place, things that help and get in the way of putting the program into place, and how the program can be scaled up to reach even more churches. The investigators will also examine the effect of the program (pre- to post-changes) on walking group member outcomes (physical activity and social cohesion). The investigators expect to work with approximately 26 AME churches for this study.

DETAILED DESCRIPTION:
Physical activity (PA) plays a critical role in preventing and treating chronic disease and promoting quality of life across the age spectrum. Older adults are a priority population for increasing PA as they experience disproportionate rates of chronic disease, are underactive, and their proportion of the US population is increasing. The proposed study, which serves as the core research project for the University of South Carolina Prevention Research Center, uses a within-site pre-post study design (i.e., quasi-experimental) to study the implementation of Walk Your Heart to Health (WYHH) by AME Churches. Churches will also receive training in how to modify organizational practices to support physical activity. The study's primary focus is to study implementation outcomes. The Consolidated Framework for Implementation Research will help inform three primary questions: (1) how do contextual factors influence implementation and sustainability success or failure? (2) what barriers and facilitators to implementation exist? and (3) how can the EBI be scaled up to broader regions or populations outside the research community? Data from pastors and church implementers will come from multiple sources (surveys, interviews, etc.) and time points and will be analyzed using a matrixed multiple case study approach and rapid qualitative analysis. The investigators will work with the CAB and other partners to ensure cultural relevance of intervention strategies and support materials in Year 1, pilot the implementation strategies and measurements in Year 2 (6 churches), conduct the implementation study in Years 3 and 4 (20 churches), and focus on translation and scale up activities in Year 5. A secondary focus is to study participant-level outcomes. Increasing PA in older adults is a Healthy People 2030 goal. Churches are vital but underutilized institutions for implementing EBIs that can contribute to reaching national priorities.

ELIGIBILITY:
Inclusion Criteria:

* Member of participating church (Charleston or Columbia Districts of the 7th Episcopal District of the AME church) or is in larger neighborhood and able to attend
* Aged 50 years and older
* Agrees to participate in in-person walking group sessions
* Not planning to move in the next year from a location that would make study visits difficult

Exclusion Criteria:

* No contraindications to exercise, as determined by the PAR-Q

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-09-29 (Estimated); Study Completion 2029-09-29 (Estimated)

PRIMARY OUTCOMES:
Pedometer steps | baseline, 8 weeks, 32 weeks
  Average steps per day from pedometer

SECONDARY OUTCOMES:
Modified version of Physical Activity Group Environment Questionnaire (Group Cohesion), as used in Walk Your Heart to Health effectiveness trial | 8 weeks, 32 weeks
  A 21-item self-reported survey that assesses the subscales of task cohesion (6 items, scores can range from 6 to 30), social cohesion (6 items, scores can range from 6 to 30), perception of group integration around task factors (5 items, scores can range from 5 to 25), and perception of group integration around social factors (4 items, scores can range from 4 to 20). For all subscales, higher scores indicate a greater sense of group cohesion or group integration.
Modified Version of the Physical Activity Group Environment Questionnaire (Leader Behaviors), as used in Walk Your Heart to Health effectiveness trial | 8 weeks, 32 weeks
  A 13-item self-report measure of how participants view the behaviors of their walking leaders. Possible scores can range from 13 to 65, with higher scores indicating more positive leader behaviors.
Supportive Accountability Inventory | 8 weeks, 32 weeks
  An 8-item self-report measure that assesses the degree to which the participant feels a sense of accountability to their walking group. Scores can range from 8 to 56, with higher scores indicating a greater sense of accountability to the walking group.
Health-Related Quality of Life (EuroQol 5 Dimensions 5 Levels; EQ-5D-5L) | baseline, 8 weeks, 32 weeks
  A 5-item self-reported measure that assesses the participants' ratings of quality of life in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. For each item, the participant chooses a statement (from a list of 5) that best describes them. Scores for each area range from 1 to 5 (1=no impairment; 5 = extreme impairment). Scores will be presented as the percentage of participants in each level for each dimension. A total score will also be computed. Possible scores on the scale range from 11111 (best possible score - no impairment on any of the 5 dimension) to 55555 (worse possible score - extreme impairments on all 5 dimensions). The score will be converted into a single index value based on country-specific norms.
Self-Efficacy for Exercise Scale | baseline, 8 weeks, 32 weeks
  A 7-item modified self-report scale in whcih participants report confidence in their ability to overcome barriers to walking 3 times per week for 50 minutes each time. Each item is rated from 0 (not confident) to 10 (very confident). Items are summed and divided by 7 so that the total score can range from 0 to 10, with higher scores indicating greater self-efficacy to overcome barriers to walking.
The UCLA 3-Item Loneliness Scale | baseline, 8 weeks, 32 weeks
  A 3-item measure that assesses 3 dimension of loneliness: relational connectedness, social connectedness, and perceived isolation. For each item, participants rate how often they experience each dimension ranging from 1 (hardly ever), to 2 (some of the time), to 3 (often). Total scores can range from 3 to 9, with higher scores indicating greater loneliness. Participants who score 3-5 are typically considered "not lonely" whereas those who score 6 to 9 are typically considered "lonely."
Church practices and policies | baseline, 8 weeks, 32 weeks
  An 11-item self-report scale used in the investigator's previous studies. Participants report how often there are opportunities, messages, and pastor support for physical activity at their church as well as the presence of policies that support physical activity. Scores for each dimension are created ranging from 1 to 4 (higher scores indicate more favorable practices/policies). A composite score which is the average of the four dimensions is also created, ranging from 1 to 4, interpreted the same way.
Self-Reported Physical Activity | baseline, 8 weeks, 32 weeks
  Participants are asked whether, in a usual week not including time at work, they do moderate or vigorous physical activity (yes or no), and if yes, how many days and how much total time per day. For those who report they do some physical activity, the investigators multiple days by time to get minutes per week of physical activity. Investigators then clasify participants as inactive (report no physical activity), underactive (report less than 150 minutes per week of physical activity), or regularly active (report 150 minutes or more per week of physical activity). The items are based on the Behavioral Risk Factor Surveillance System questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Wilcox, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Free public access to de-identified participant data will be provided within 30 months of completion of the project. Data will include all primary and secondary outcomes along with basic descriptive information.
Supporting Information: Analytic Code
Time Frame: Free public access to de-identified participant data will be provided within 30 months of completion of the project. The investigators will use an external housing source to keep data available from the site.
Access Criteria: Free, open source access.